CLINICAL TRIAL: NCT04777747
Title: The Role of Lactate From Viral to Bacterial Infection
Brief Title: The Role of Lactate in Viral and Bacterial Infection
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Children's Hospital of Chongqing Medical University
Other Study IDs: lactate for infection
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-10

CONDITIONS: Viral Infection; Bacterial Infections; Lactate Blood Increase
MeSH Terms: conditions — Virus Diseases; Bacterial Infections; Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- viral infection: a child is infected by virus only
  Interventions: Other: viral infection
- viral and bacterial infection: a child is infected by virus and progress to bacterial infection
  Interventions: Other: viral and bacterial infection

INTERVENTIONS:
Other: viral infection — a child is infected by virus only
  Groups: viral infection
Other: viral and bacterial infection — a child is infected by virus and progress to bacterial infection
  Groups: viral and bacterial infection

SUMMARY:
Acute upper respiratory tract infection(AURI) is common in children, and viral infection is the main cause. However, several children with viral infection are easy to suffer from secondary bacterial infection, and the mechanism is unclear.

DETAILED DESCRIPTION:
Lactate is an important molecule in the spread and metastasis of tumor by suppressing the innate immune response. As is known, the immune system is not mature in children and it is reverse related to the age of children. An reasonable hypothesis is that the lactate is a independent risk factor in the children with viral infection progress to bacterial infection. Here, our aim is to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* child's age is from 0 to 18 years
* a child is at least diagnosed with viral infection

Exclusion Criteria:

one of the following conditions appeared:

* congenital heart disease or other abnormalities
* respiratory failure
* hereditary and/or metabolic disease

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The age of a child ranged from 0 to 18 is included in the present study, especially the first viral infection.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
level of lactate | three days after admission
  level of lactate in both viral and viral and bacterial infection groups
the level of lactate dehydrogenase(LDH) | three days after admission
  level of LDH in both viral and viral and bacterial infection groups

CONTACTS AND LOCATIONS:
Locations (1):
- Chen, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
two years after the study accomplishment
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from Jan-1, 2025 to Dec-31, 2025